CLINICAL TRIAL: NCT05864235
Title: Texting to Reduce Alcohol Misuse Pilot Trial
Acronym: TRAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brian Suffoletto, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 67584
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Consumption
Keywords: young adults; binge drinking; text message
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Each week for 6-weeks, control group participants will receive the following weekly text message assessments (without receiving any feedback or support): (1) Thursdays (3pm): weekend plans to drink and desire to get drunk; (2) Sundays (12pm): most drinks consumed on any weekend day and peer pressure to drink.
  Interventions: Behavioral: Control
- Goal Support (GS) (Experimental): Each week for 6-weeks, GS group participants will compete identical weekly text message assessments to the control group and receive further prompts and tailored feedback and support focused on weekly drinking limit goal commitment & confidence assessments and subsequently receive tailored feedback on goal success to either bolster future goal striving or reframe goal failure.
  Interventions: Behavioral: Control; Behavioral: Goal Support (GS)
- GS + Coaching for Context-specific Peer Support (CCPS) (Experimental): Each week for 6-weeks, CCPS group participants will compete identical weekly text message assessments and feedback to GS plus additionally will receive weekly motivation and strategies to enlist peer support during drinking episodes.
  Interventions: Behavioral: Control; Behavioral: Goal Support (GS); Behavioral: Coaching for Context-specific Peer Support (CCPS)

INTERVENTIONS:
Behavioral: Control — Each week for 6-weeks, control group participants will receive the following weekly text message assessments (without receiving any feedback or support): (1) Thursdays (3pm): weekend plans to drink and desire to get drunk; (2) Sundays (12pm): most drinks consumed on any weekend day and peer pressure to drink.
Behavioral: Goal Support (GS) — Each week for 6-weeks, GS group participants will receive prompts and tailored feedback and support focused on weekly drinking limit goal commitment & confidence assessments and subsequently receive tailored feedback on goal success to either bolster future goal striving or reframe goal failure.
  Arms: GS + Coaching for Context-specific Peer Support (CCPS); Goal Support (GS)
Behavioral: Coaching for Context-specific Peer Support (CCPS) — Each week for 6-weeks, CCPS group participants will receive weekly motivation and strategies to enlist peer support during drinking episodes.
  Arms: GS + Coaching for Context-specific Peer Support (CCPS)

SUMMARY:
The primary aims of this project are to determine the feasibility and acceptability of recruiting and retaining young adult binge drinkers online and using text messaging to provide weekly Goal Support (GS) or weekly GS + Coaching for Context-specific Peer Support (CCPS) on alcohol consumption. The secondary aims will determine effect sizes for GS and GS+CCPS groups relative to controls on alcohol consumption at 6- and 12-weeks to inform design of an adequately-powered trial.

ELIGIBILITY:
Inclusion Criteria:

* English reader
* Owns a mobile phone with SMS
* Hazardous alcohol consumption as measured by: "How many times in the past year have you had X or more drinks in a day?", where X is 5 for men and 4 for women, and a response of 1 or greater is considered at-risk
* At least in contemplative stage of change for reducing alcohol consumption

Exclusion Criteria:

* Currently enrolled or past enrollment in a 4-year college
* Pregnant or pregnancy plans in the next 3-months
* Current or planned treatment for alcohol or substance use disorder in next 3-months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The % of people screened to participants enrolled | 2 months
  Online recruitment efficiency
The % of participants who complete both 6- and 12-week web-based assessments | 12 weeks
  Follow-up completion
The % of SMS queries with valid responses | 6 weeks
  Response rates to SMS queries
The % of participants who at least agree that the SMS program helped them reduce their drinking | 12 weeks
  A single question with response options: completely disagree to completely agree

SECONDARY OUTCOMES:
# Binge drinking days | 6-weeks
  Count of binge drinking days using TLFB 30-day calendar
Binge drinking days | 12-weeks
  Count of binge drinking days using TLFB 30-day calendar
Drinks per drinking day | 6-weeks
  Mean drinks per drinking day using TLFB 30-day calendar
Drinks per drinking day | 12-weeks
  Mean drinks per drinking day using TLFB 30-day calendar
# Alcohol negative consequences | 6-weeks
  B-YAACQ: 24 yes/no questions
Alcohol negative consequences | 12-weeks
  B-YAACQ: 24 yes/no questions

CONTACTS AND LOCATIONS:
Overall Officials: Brian Suffoletto, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States